CLINICAL TRIAL: NCT04817111
Title: A Phase 2a Study of NAD+ Precursor Supplementation in Friedreich's Ataxia
Brief Title: NAD+ Precursor Supplementation in Friedreich's Ataxia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Metro International Biotech, LLC (Industry)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Shana McCormack, Attending Physician, Children's Hospital of Philadelphia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19-016525; MIB-626-201 (Other: Metro International Biotech, LLC)
Record Dates: First submitted 2021-03-10; First posted 2021-03-25 (Actual); Results first posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Friedreich Ataxia
MeSH Terms: conditions — Friedreich Ataxia

STUDY DESIGN:
Intervention Model Description: Open Label, 14 Days (+/- 2 Days)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label - MIB-626 (Other): MIB-626
  Interventions: Drug: MIB-626

INTERVENTIONS:
Drug: MIB-626 — Two (2) 500 mg Tablets, By Mouth, Daily

SUMMARY:
The primary objective is to test the safety and tolerability of short-term therapy with a nicotinamide adenine dinucleotide (NAD+) precursor (MIB-626) in adults with Friedreich's Ataxia (FA) without overt heart failure and with a left ventricular ejection fraction ≥ 40%. A key secondary objective is to test the effects of MIB-626 on cardiac and skeletal muscle bioenergetics.

DETAILED DESCRIPTION:
The primary focus for this protocol is safety and tolerability. We will systematically assess for adverse events using a safety monitoring uniform report form. We will also use cardiac 31-Phosphorus-Magnetic Resonance Spectroscopy (MRS) to measure the Phosphocreatine(PCr)/Adenosine triphosphate (ATP)- γ ratio before and after treatment with MIB-626. In addition, if time permits we will use proton (1H)-MRS to measure skeletal muscle nicotinamide adenine dinucleotide (NAD+) before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Molecular diagnosis of Friedreich's Ataxia (FA).
* Males and females, ages 18 years to < 65 years.

Exclusion Criteria:

* Known sensitivity to nicotinamide-containing compounds.
* Concurrent use of Vitamin B3 supplements and/or any medications likely to increase risk of MIB-626 toxicity.
* HgbA1c > (great than or equal to) 8.5% and or Diabetes Mellitus (DM) requiring insulin or insulin secretagogue.
* Kidney disease (Estimated Glomerular Filtration Rate (eGFR) < 60 ml/min/1.73 m2) using serum creatinine and MDRD equation. The eGFR levels will be calculated using the Modified Diet in Renal Disease Study (MDRD) equation, which is the equation used by the Children's Hospital Of Philadelphia laboratory.
* Liver disease (Aspartate Aminotransferase (AST)/Alanine Aminotransferase (ALT) > 3 x Upper Limit of Normal)
* Severe co-existing cardiac disease (Ejection Fraction (EF) < 40%, known arrhythmia) as demonstrated by an echocardiogram within 12 months of screening.
* Any contraindication to MRI, including spinal rods (related to unknown safety considerations for cardiac 31-Phosphorus -MRS).
* Use of any investigational agent within 4 weeks of enrollment.
* Females: Pregnant/lactating or planning to become pregnant during their participation.
* Any medical condition that, in the opinion of the investigator, will interfere with the safe completion of the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2022-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shana E McCormack, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
IPD may be available with appropriate regulatory approvals.

REFERENCES:
- [Background] DeBrosse C, Nanga RPR, Wilson N, D'Aquilla K, Elliott M, Hariharan H, Yan F, Wade K, Nguyen S, Worsley D, Parris-Skeete C, McCormick E, Xiao R, Cunningham ZZ, Fishbein L, Nathanson KL, Lynch DR, Stallings VA, Yudkoff M, Falk MJ, Reddy R, McCormack SE. Muscle oxidative phosphorylation quantitation using creatine chemical exchange saturation transfer (CrCEST) MRI in mitochondrial disorders. JCI Insight. 2016 Nov 3;1(18):e88207. doi: 10.1172/jci.insight.88207. PMID 27812541
- [Background] Bagga P, Wilson N., DeBrosse D., Hariharan H., Reddy R., editor. In vivo detection of NAD+ in human calf muscle at 7T using 28-channel knee volume coil. International Society for Magnetic Resonance in Medicine; 2019; Montreal, Canada.
- [Background] Patel M, Isaacs CJ, Seyer L, Brigatti K, Gelbard S, Strawser C, Foerster D, Shinnick J, Schadt K, Yiu EM, Delatycki MB, Perlman S, Wilmot GR, Zesiewicz T, Mathews K, Gomez CM, Yoon G, Subramony SH, Brocht A, Farmer J, Lynch DR. Progression of Friedreich ataxia: quantitative characterization over 5 years. Ann Clin Transl Neurol. 2016 Jul 25;3(9):684-94. doi: 10.1002/acn3.332. eCollection 2016 Sep. PMID 27648458

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Open Label - MIB-626
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Open Label - MIB-626
Number analyzed (Participants) | 7
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 26 [26 to 33.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Individuals With Treatment-emergent Adverse Events as Assessed by Common Terminology Criteria for Adverse Events Version 5.0.
Description: Safety will be monitored through collection of laboratory assessments (CBC, complete metabolic profile, lipid profile, HbA1c), vital signs (heart rate, blood pressure), and ECG, all of which will be reviewed for clinically relevant abnormalities, and standardized assessment of symptoms. We report the proportion of individuals who had at least one treatment-emergent adverse event of Grade 1 or higher.
Time Frame: 14 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label - MIB-626
Number analyzed (Participants) | 7
Participants | 4

2. Secondary Outcome: Cardiac 31-Phosphorus-Magnetic Resonance Spectroscopy (MRS): Phosphocreatine (PCr)/Adenosine Tri-Phosphate (ATP) Ratio
Description: Measure the within-participant change in PCr/ATP ratio before and after treatment with MIB-626.
Time Frame: Change from baseline to 14 days.
Population: 1/7 individuals was unable to complete an MRI scan.
Measure: Median (Inter-Quartile Range); unit: PCr to ATP ratio
Arm/Group | Open Label - MIB-626
Number analyzed (Participants) | 6
PCr to ATP ratio | -0.445 [-0.6025 to -0.0925]
Statistical Analysis 1: Comparison: Open Label - MIB-626; Test type: Other — Wilcoxon signed-rank test was used to test if the change from pre- vs. post-test outcome is different from zero; p = 0.18, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Post-Exercise Creatine Chemical Exchange Saturation Transfer (CrCEST) Magnetic Resonance Imaging (MRI)
Description: Assess the within-participant change in skeletal muscle post-exercise CrCEST recovery (an index of skeletal muscle mitochondrial oxidative phosphorylation capacity).
Time Frame: Change from baseline to 14 days.
Population: This secondary outcome measure could not be collected for any participant because insufficient MRI scanning time remained during the visits after main outcomes were collected.
Arm/Group | Open Label - MIB-626
Number analyzed (Participants) | 0

4. Secondary Outcome: Grip Strength
Description: Assess within-participant changes in grip strength (via hand grip dynamometry) before and after treatment with MIB-626.
Time Frame: Change from baseline to 14 days.
Measure: Median (Inter-Quartile Range); unit: kg
Arm/Group | Open Label - MIB-626
Number analyzed (Participants) | 7
kg | -0.65 [-2.625 to -0.075]
Statistical Analysis 1: Comparison: Open Label - MIB-626; Test type: Other — Wilcoxon signed-rank test was used to test if the change from pre- vs. post-test outcome is different from zero; p = 0.21, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Concentration of Nicotinamide Adenine Dinucleotide (NAD+) in Whole Blood
Description: Measure the concentration of NAD+ in whole blood before and after treatment with MIB-626.
Time Frame: Change from baseline to 14 days.
Measure: Median (Inter-Quartile Range); unit: micro-molar
Arm/Group | Open Label - MIB-626
Number analyzed (Participants) | 6
micro-molar | 49.9 [42 to 54]
Statistical Analysis 1: Comparison: Open Label - MIB-626; Test type: Other — Wilcoxon signed-rank test was used to test if the change from pre- vs. post-test outcome is different from zero; p = 0.03, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | Open Label - MIB-626
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 4/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label - MIB-626 (N=7)
Belching (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2022-05-06): https://cdn.clinicaltrials.gov/large-docs/11/NCT04817111/Prot_003.pdf
  • Statistical Analysis Plan (2022-05-06): https://cdn.clinicaltrials.gov/large-docs/11/NCT04817111/SAP_004.pdf
  • Informed Consent Form (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/11/NCT04817111/ICF_000.pdf